CLINICAL TRIAL: NCT05775861
Title: Dexmedetomidine Added to Ropivacaine Single Shot vs Continuous Interscalene Nerve Block for Elective Arthroscopic Shoulder Surgery: a Prospective Randomized Control Trial
Brief Title: Dexmedetomidine Added to Ropivacaine Single Shot vs Continuous Interscalene Nerve Block
Acronym: DEXBIB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Ariane Clairoux, MD, Assistant professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2892
Record Dates: First submitted 2023-01-03; First posted 2023-03-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia; Shoulder Pain; Post Operative Pain
Keywords: Dexmedetomidine; interscalene brachial plexus nerve blocks; Elective ambulatory minor shoulder surgery
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: All patients will be first met either at our preoperative investigation clinic or by phone in the days leading to surgery to present the project and obtain consent. Consent will be dynamic and participants will have the possibility to withdraw from the study at all times.
  A web-based inclusion and randomization form will be provided to the investigators. Randomization will be done in a 1:1 ratio. Envelopes will be made, one for each patient, and will contain the randomization information and in which group they are in: D in the single shot dexmedetomidine added to ropivacaine or R for the continuous interscalene brachial plexus block with ropivacaine.
Masking Description: The patient, the anesthesiologist that will perform the block and the operating room staff cannot be blinded for treatment group allocation since the material differs in the 2 groups. We did not want to remain blind at all costs by installing catheters in all participants, with a continuous infusion of saline for the dexmedetomidine group, since the insertion of a catheter is not without risk for the patient and the initial bolus would have been diluted.
  The nurse staff, anesthesiologists and the research staff evaluating the patient by phone on postoperative days 1,2 and 3 will not be blinded to the patients' study care group allocation because they will also be looking for minor complications that involve the catheter or the infusion pump.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single shot interscalene brachial plexus with dexmedetomidine added to ropivacaine (Experimental): A total of 150 mg of ropivacaine 0.5% will be prepared, 125 mg (25mL) will be mixed with a dose of 2 mcg/kg IBW of dexmedetomidine (100 mcg/mL dexmedetomidine hydrochloride; Precedex, Hospira Inc, Lake Forest, IL). The total of 25 mL (125 mg or ropivacaine 0.5%) with dexmedetomidine will be injected perineurally at the level of the roots and a 5 mL (25 mg) will be injected between the sternocleidomastoid muscle and anterior scalene for the superficial cervical plexus block.
  Interventions: Drug: single shot interscalene brachial plexus block group with dexmedetomidine added to ropivacaine group
- continuous interscalene brachial plexus block with ropivacaine (Active Comparator): A total of 100 mg (20 mL) of ropivacaine 0,5% will be injected perineurally at the level of the roots using the Tuohy needle. The 19 G arrow catheter will then be introduced through the Tuohy needle and we will leave 4 cm of the catheter perineurally. An additional 25 mg (5 mL) of ropivacaine 0,5% will be injected using the catheter to make sure the catheter is in a correct position. An additional 5 mL (25 mg) of ropivacaine 0.5 % will be injected between the sternocleidomastoid muscle and anterior scalene for the superficial cervical plexus block using an ultrasound in-plane approach with a 22 G 80-mm ultrasound needle (Pajunk SonoTAP II, Germany) or with a standard 25G 1 1/2 inches needle. After the surgery, an infusion of ropivacaine 0,2% at a standard rate of 5 mL/h will be started using an elastomeric pump of 300 mL (Baxter Corporation, Mississauga, Ontario).
  Interventions: Drug: continuous interscalene brachial plexus block

INTERVENTIONS:
Drug: single shot interscalene brachial plexus block group with dexmedetomidine added to ropivacaine group — For the single shot group with dexmedetomidine added to ropivacaine group (Group D), after local analgesia with 3 mL of 1% lidocaine, the block will be performed under ultrasound guidance using an in-plane approach with a 22 G 80-mm ultrasound needle (Pajunk SonoTAP II, Germany).
  The perineural solution will be pre-mixed in a 30 mL syringe before the realization of the block.
  A total of 150 mg of ropivacaine 0.5% will be prepared, 125 mg (25mL) will be mixed with a dose of 2 mcg/kg IBW of dexmedetomidine (100 mcg/mL dexmedetomidine hydrochloride; Precedex, Hospira Inc, Lake Forest, IL). The total of 25 mL (125 mg or ropivacaine 0.5%) with dexmedetomidine will be injected perineurally at the level of the roots and a 5 mL (25 mg) will be injected between the sternocleidomastoid muscle and anterior scalene for the superficial cervical plexus block.
  Arms: single shot interscalene brachial plexus with dexmedetomidine added to ropivacaine
Drug: continuous interscalene brachial plexus block — The block will be performed under ultrasound guidance using an in-plane approach with a 17G Tuohy needle (Arrow FlexBlock). A total of 100 mg (20 mL) of ropivacaine 0,5% will be injected perineurally at the level of the roots using the Tuohy needle. The 19 G arrow catheter will then be introduced through the Tuohy needle and we will leave 4 cm of the catheter perineurally. An additional 25 mg (5 mL) of ropivacaine 0,5% will be injected using the catheter to make sure the catheter is in a correct position. An additional 5 mL (25 mg) of ropivacaine 0.5 % will be injected between the sternocleidomastoid muscle and anterior scalene for the superficial cervical plexus block using an ultrasound in-plane approach with a 22 G 80-mm ultrasound needle (Pajunk SonoTAP II, Germany) or with a standard 25G 1 1/2 inches needle. After the surgery, an infusion of ropivacaine 0,2% at a standard rate of 5 mL/h will be started using an elastomeric pump of 300 mL (Baxter Corporation, Mississauga, Ontario).
  Arms: continuous interscalene brachial plexus block with ropivacaine

SUMMARY:
Arthroscopic shoulder surgery is increasingly performed in an outpatient setting and post-operative pain management is often a real challenge as those surgeries are well recognized for their high level of pain which often affects physical rehabilitation. The interscalene block is a largely used anesthetic technique to perform these surgeries whilst avoiding general anesthesia (GA) and to provide postoperative analgesia. However, the painful period often exceeds the duration of a single shot block, thus affecting patient recovery. Some specialized centers use a continuous catheter and elastomeric pump in order to prolong the duration of analgesia. However, several logistical, professional and financial constraints limit the use of these catheters and pumps in a great number of outpatient centers. On the other hand, perineural dexmedetomidine is increasingly used as an adjuvant to improve block onset, analgesia duration and patient satisfaction.

The use of adjuvants such as perineural dexmedetomidine added to a single shot interscalene block appears to be an interesting option to prolong postoperative analgesia without the limitations imposed by a continuous catheter and elastomeric pumps in arthroscopic shoulder surgeries.

DETAILED DESCRIPTION:
A growing number of arthroscopic shoulder surgeries are performed in an ambulatory setting. For these patients, postoperative pain management is an important factor for analgesia and optimal rehabilitation. Peripheral nerve blocks, and more particularly the interscalene brachial plexus block (ISB), is the method of choice to provide adequate surgical conditions and satisfactory postoperative pain control for shoulder surgeries. Even before the advent of ultrasound guidance , interscalene blocks resulted in a high level of patient satisfaction, fewer post-operative complications and a reduction of hospital stay compared to general anesthesia.

Shoulder surgeries are well recognized to cause severe postoperative pain, mainly in the first 48h, and the use of a single shot interscalene block (SSISB) is limited by its duration of action, which often fails to cover the duration of postoperative analgesia beyond 24 hours.

On the other hand, ultrasound-guided continuous interscalene blocks (CISB) have shown a significant reduction of pain compared to single shot interscalene blocks. However, CISB are limited by many logistical problems which make their use difficult in most ambulatory centers. Indeed, catheter placement is often a technically challenging procedure and accidental catheter removal is a complication that limits their usefulness. However, when the necessary technical resources and medical expertise is available, CISB have been associated with a superior level of analgesia, reduction of opioid consumption, improvements in rest and dynamic pain, and lower instances of postoperative nausea and vomiting than SSISB in major shoulder surgery. A recent study has demonstrated that automated intermittent boluses did not provide better analgesia nor reduced rescue opioid consumption compared to continuous infusion of ropivacaine despite both groups describing insufficient pain relief.

The persistence of pain despite the use of SSISB or CISB has lead several anesthesia teams to use adjuvants to improve the effect and duration of analgesia. Over the years, several adjuvants have been administered to enhance the brachial plexus block onset and duration. Thus, intravenous dexamethasone administered at the time of performing ISB is widely used to improve the duration of analgesia following shoulder surgeries. In addition to the benefits already provided by the addition of intravenous dexamethasone, there is also an added value to perineural dexmedetomidine in order to accelerate the onset of motor and sensory block, extend the duration of the block and reduce the pain score 14 hours postoperatively in elective shoulder surgery.

The combination of intravenous or perineural dexmedetomidine, an α-2 adrenoceptor agonist, with ropivacaine prolongs the duration of SSISB analgesia and reduces opioid consumption postoperatively without prolonging the duration of motor blockade during outpatient shoulder surgeries. Patients undergoing elective shoulder surgery under general anesthesia with perineural dexmedetomidine added to ropivacaine for interscalene block had a faster sensory and motor block onset, an increased duration of nerve blockade and improved postoperative pain up to 14h after the block. Even when a peripheral nerve block is used as the primary anesthetic, SSISB with perineural dexmedetomidine added to ropivacaine in arthroscopic rotator cuff repair has shown lower pain and improved patient satisfaction within 48 h postoperatively. The perfect perineural dexmedetomidine dose should provide optimal analgesia with minimal side effects such as hypotension and bradycardia. Over the years, it has been used in wide-ranging doses and 2 mcg/kg seems to be the optimal dose in SSISB for arthroscopic shoulder surgery to obtain a suitable duration of analgesia. A recent meta-analysis demonstrates the safety of perineural dexmedetomidine as well as its effectiveness during brachial plexus block to accelerate the onset of action and prolong the duration of analgesia. Indeed, no neurological complications or neurotoxic symptoms were reported in patients who received perineural dexmedetomidine.

Rationale for this study:

The addition of dexmedetomidine to ropivacaine for SSIB could improve the duration of postoperative analgesia and patient satisfaction for arthroscopic shoulder surgeries without the limitations and potential complications of an CISB catheter and elastomeric pump. Moreover, the use of a catheter is a complex procedure compared to a single injection and thus limited in some centers due to logistical limitations. Therefore, SSISB with perineural dexmedetomidine could be an interesting alternative to perform shoulder surgeries in centers where the use of a continuous catheter is limited by technical, professional or financial resources. Ultimately, this improvement in postoperative analgesia could lead to early patient mobilization, better physical rehabilitation and improved patient satisfaction. This study will focus on recovery, to better understand patient outcomes and experiences as a whole, in this era of personalized medicine and patient oriented research.

Methods: A predetermined sample size of patients of more than18 years old, ASA status I-III scheduled to undergo elective minor ambulatory shoulder surgery are included. Patients with known allergy to local anesthetics, contraindication to interscalene brachial plexus nerve block or superficial cervical plexus block will be excluded. The premedication and peripheral nerve block technique will be standardized for both groups. Patients will be randomized to receive either a single shot interscalene block with 150 mg of isobaric ropivacaine 0.5% (125 mg at the interscalene brachial plexus level and 25 mg at the superficial cervical plexus) with 2 mcg/kg (IBW) of dexmedetomidine or a continuous interscalene block with an initial dose of 150 mg of isobaric ropivacaine 0.5% (125 mg at the interscalene brachial plexus level and 25 mg at the superficial cervical plexus) and an infusion using an elastomeric pump of 300 mL at a rate of 5 mL/h of isobaric ropivacaine 0.2% for 60 hours. The primary endpoint will be the Quality of Recovery (QoR-15) questionnaire at 48h. The secondary endpoints will be: QoR-15 at 24h and 72h, time before the first analgesic request, time before the end of sensory block, time before the end of motor block, patient satisfaction, total post-operative opioid consumption, major and minor complications.

Study design: Prospective, randomized controlled trial.

Subject population: Adult patients scheduled to undergo elective arthroscopic ambulatory shoulder surgery

Sample size: 96

Study duration: 12 months

Study center: CIUSSS de l'Est de l'Ile de Montréal, Montreal, QC, Canada

Adverse Events: None expected

Subvention: applications to the Canadian Society of Anesthesia as well as to the Foundation of the Association of the Anesthesiologists of Quebec and to the department of anesthesiology of the UdeM will be proposed within the coming year 2021-2022.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* ASA status of I-III
* Patients undergoing elective arthroscopic ambulatory shoulder surgery
* Anticipated return home the same day (less than 12 hours in-hospital) in any operating theater of the CIUSSS.

Exclusion Criteria:

* less than 18 years old
* Patient refusal
* Pregnancy
* Patients with known allergy to local anesthetics
* Contraindication to interscalene brachial plexus nerve block or superficial cervical plexus block: coagulopathy, contralateral phrenic nerve dysfunction, infection at the puncture site, severe chronic obstructive pulmonary disease
* Technical inability to proceed with the interscalene brachial plexus nerve block
* Surgery requiring general anesthesia
* Body weight less than 50 kg
* Patient with no family member or caring adult at home during the first 72h postoperative (contraindication to elastomeric pump)
* Unable to communicate with the investigators, unable to read the questionnaire, unable to keep track and notes of the medication taken at home
* Significant psychiatric or cognitive condition interfering with the ability to provide consent or assessment
* Preexisting neurologic deficits or neuropathy affecting the brachial plexus
* Any contra-indication to same-day surgery identified by the pre-operative clinic such as, but not limited to, any cognitive disorder, any physical limitation other than the one leading to surgery that might impair the patient to take care of himself/herself at home, any severe pulmonary or cardiac disorder, bleeding disorder, etc,
* Any cardiac or pulmonary condition that precludes the risk of bradycardia or hypotension such as but not limited to symptomatic coronary disease, severe aortic stenosis, moderate to severe pulmonary hypertension, congestive heart failure, second or third degree block, pre-existing bradycardia (HR lower than 50), pre-existing hypotension (SBP lower than 100 mmHg), etc.
* History of chronic pain with daily opioid use during the 3 months before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint will be the Quality of Recovery (QoR-15) questionnaire score from minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery) at 48 hours postoperative. | 72 hours
  To compare the QoR-15 questionnaire scores at 48 hours postoperative after an elective arthroscopic ambulatory shoulder surgery done solely under interscalene block and superficial cervical plexus block with a single shot of 150 mg isobaric ropivacaine 0.5% with 2 mcg/kg (IBW) of dexmedetomidine (125 mg at the level of the interscalene brachial plexus and 25 mg at the level of the superficial cervical plexus) versus a continuous interscalene brachial plexus block with an initial dose of 150 mg of isobaric ropivacaine 0.5% (125 mg at the interscalene brachial plexus level and 25 mg at the superficial cervical plexus) and a continuous infusion using an infusion pump of 300 mL at a rate of 5 mL/h of isobaric ropivacaine 0.2% for 60 hours. Assessment will be done preoperatively and on postoperative day 1, day 2 (for the primary outcome) and also on day 3.

SECONDARY OUTCOMES:
QoR-15 at 24 hours and 72 hours | 24 hours and 72 hours
  To compare the Quality of Recovery-15 (QoR-15) questionnaire scores at 24 hours and 72 hours postoperative from minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).
Time before the first analgesic request | From immediate postoperative period to 72 hours postoperative
  This is defined as the time (minutes) between the ISB and the first need for rescue analgesic.
Time before the end of sensory block | From immediate postoperative period to 72 hours postoperative
  This is defined as the time (minutes) between the ISB and the time the participant felt that their shoulder sensory had return to normal.
Time before the end of motor block | From immediate postoperative period to 72 hours postoperative
  This will be defined as the time (minutes) between the ISB and the time the participant regains function of the biceps strength. Biceps strength is selected in lieu of shoulder abduction, as postoperative bandaging and the sling precludes this motion.
Patient satisfaction | 72 hours
  Patient satisfaction will be noted on a scale of 0 (poor) to 10 (excellent). Since the QoR-15 is a questionnaire comprising scales ranging from 0 to 10, we opted to assess the overall patient satisfaction on a scale of 0 to 10, 0 being completely dissatisfied and 10 being completely satisfied. We evaluate the global satisfaction on post-operative day 3 (at 72 hours postoperative).
Total post-operative opioid consumption | 72 hours
  Defined as the total equivalent of oral morphine taken during the first 3 post-operative days. Opioid consumption in the PACU will also be recorded.
Incidence of side effects related to dexmedetomidine in PACU: hypotension | 6 hours
  Hypotension will be defined as a mean arterial pressure (MAP) under 60 mmHg
Incidence of side effects related to dexmedetomidine in PACU: bradycardia. | 6 hours
  Bradycardia will be defined as a frequency cardiac (FC) under 50 beats per minute (bpm).
Major and minor complications | 72 hours
  Major complications are defined as requiring significant additional medical or surgical intervention or hospitalization. Minor complications require only observation and include: leaking catheter, early catheter withdrawal, catheter site drainage, pump leaking, hematoma, pain at the catheter site, dysphagia, hoarseness, dizziness, rash, paresthesia in the distal extremity.
Total time from end of surgery to obtention of discharge criterias. | From immediate postoperative period to 5 hours postoperative
  Total time from end of surgery to obtention of discharge criterias.
The presence of nausea and vomiting in the PACU and during the first three post-operative days. | 72 hours
  The presence of nausea and vomiting in the PACU and during the first three post-operative days.
Standardized intraoperative opioid consumption (mcg of fentanyl) | Surgery period (intraoperative)
  Standardized intraoperative opioid consumption (mcg of fentanyl)
Standardized intraoperative ketamine consumption (mg) | Surgery period (intraoperative)
  Intraoperative ketamine in mg
Standardized intraoperative total dose of propofol used for sedation (mg). | Surgery period (intraoperative)
  intraoperative total dose of propofol used for sedation (mg).

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Clairoux, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada